CLINICAL TRIAL: NCT05822349
Title: Impact of Using Pictograms as an Educational Strategy on Improving Patient Depression and Anxiety Among Low Health Literate Patients With Type 2 Diabetes at Northern Badya Hospital, Jordan.
Brief Title: Effect of Using Pictograms on Improving Depression and Anxiety Among Type 2 Diabetic Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Esraa AL Sbaihat, postgraduated student, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MOH/REC/2022/411
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): they will receive the usual diabetes care routine plus a pictogram-enriched label.
  Interventions: Behavioral: picograms-enriched label
- control group (Placebo Comparator): they will receive the usual diabetes care routine.
  Interventions: Behavioral: picograms-enriched label

INTERVENTIONS:
Behavioral: picograms-enriched label — The intervention care includes usual care (instructions for using each anti-diabetic drug) plus pictograms that show how much medications should be taken at each time of day (morning, noon, evening, and night), how to take them in relation to meals, the purpose of the drug, and the most important non-pharmacologic interventions for diabetic patients (weight loss, exercise, avoiding smoking, blood sugar controlling).

SUMMARY:
we will study the impact of using pictograms on improving depression and anxiety among type 2 diabetic patients, we suppose that patients who received pictograms-enriched labels will have lower levels of depression and anxiety in comparison with those who will not receive after three month follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible if they are Jordanian adults, aged 18 or older, who have been clinically diagnosed with T2DM for at least 6 months, having low health literacy (Individuals who obtained 66 or lower scores in the full TOFHLA instrument are considered as individuals with "low literacy" in the study) [24], come personally for the refill.

Exclusion Criteria:

* Patients who are unable to communicate verbally (aphasic or with hearing impairment), those with any visual, learning disabilities, and psychological or hepatorenal disease (according to the clinical diagnosis by a physician), and those deemed too ill or frail to attend the clinic, and who have participated in other diabetes education research projects will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
change in depression level | 12 weeks following ends of intervention
  Patient Health Questionnaire-9 (PHQ-9)
change in anxiety level | 12 weeks following ends of intervention
  Generalized Anxiety Disorder scale (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: AL-Motassem F Yousef, Study Director — University of Jordan
Locations (1):
- Northern Badya Hospital, Al Mafraq, Jordan

IPD SHARING:
Plan to Share IPD: Undecided